CLINICAL TRIAL: NCT03924856
Title: A Phase 3, Randomized, Double-blind Study to Evaluate Perioperative Pembrolizumab (MK-3475) + Neoadjuvant Chemotherapy Versus Perioperative Placebo + Neoadjuvant Chemotherapy in Cisplatin-eligible Participants With Muscle-invasive Bladder Cancer (KEYNOTE-866)
Brief Title: Perioperative Pembrolizumab (MK-3475) Plus Neoadjuvant Chemotherapy Versus Perioperative Placebo Plus Neoadjuvant Chemotherapy for Cisplatin-eligible Muscle-invasive Bladder Cancer (MIBC) (MK-3475-866/KEYNOTE-866)
Acronym: KEYNOTE-866
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-866; MK-3475-866 (Other: MSD Protocol Number); KEYNOTE-866 (Other: MSD); 2080224790 (Registry Identifier: jRCT); 2022-501970-20-00 (Registry Identifier: EU CT); 194870 (Registry Identifier: JAPAC-CTI); U1111-1282-6279 (Registry Identifier: UTN); 2018-003808-39 (EudraCT Number)
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Pembrolizumab (MK-3475); Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Gemcitabine; Cisplatin; Surgical Procedures, Operative; Cystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Gemcitabine + Cisplatin + Surgery (Experimental): Participants received 4 preoperative cycles of pembrolizumab PLUS gemcitabine PLUS cisplatin, followed by surgery, followed by up to 13 cycles of postoperative pembrolizumab.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin; Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND])
- Placebo + Gemcitabine + Cisplatin + Surgery (Placebo Comparator): Participants received 4 preoperative cycles of placebo to pembrolizumab PLUS gemcitabine PLUS cisplatin, followed by surgery, followed by up to 13 cycles of postoperative placebo to pembrolizumab.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND]); Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg by intravenous (IV) infusion, given on Day 1 of each 21-day cycle
  Other Names: MK-3475
  Arms: Pembrolizumab + Gemcitabine + Cisplatin + Surgery
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2, IV infusion on Days 1 and 8 of each 21-day cycle
Drug: Cisplatin — Cisplatin 70 mg/m^2, IV infusion on Day 1 of each 21-day cycle
Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND]) — Surgical RC+PLND will be done in accordance with the American Urological Association (AUA)/American Society of Clinical Oncology (ASCO)/American Society for Radiation Oncology (ASTRO)/Society of Urologic Oncology (SUO) guidelines.
Drug: Placebo — Placebo to pembrolizumab by IV infusion, given on Day 1 of each 21-day cycle
  Arms: Placebo + Gemcitabine + Cisplatin + Surgery

SUMMARY:
A global study to evaluate peri-operative pembrolizumab with chemotherapy versus placebo to pembrolizumab plus chemotherapy in cisplatin eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of urothelial carcinoma (UC) / muscle invasive bladder cancer (MIBC) (T2-T4aN0M0 or T1-T4aN1M0) with predominant (≥50%) urothelial histology.
* Have clinically non-metastatic bladder cancer (N≤1 M0) determined by imaging (computed tomography (CT) or magnetic resonance imaging (MRI)) of the chest/abdomen/pelvis.
* Be deemed eligible for Radical Cystectomy (RC) + Pelvic Lymph Node Dissection (PLND).
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Have adequate organ function.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active anti-cancer treatment ≤3 years of study randomization with certain exceptions.
* Has received any prior systemic treatment for MIBC or non-invasive muscle bladder cancer (NMIBC - prior treatment for NMIBC with intravesical BCG/chemotherapy is permitted) or prior therapy with an anti- programmed cell death 1 (PD-1), anti-programmed cell death ligand 1/ ligand 2 (PD-L1/L2), or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4).
* Has ≥N2 disease or metastatic disease (M1) as identified by imaging.
* Is cisplatin-ineligible, as defined by meeting any one of the cisplatin ineligibility criteria as per protocol.
* Has received prior systemic anticancer therapy including investigational agents within 3 years of randomization or any radiotherapy to the bladder.
* Has undergone partial cystectomy of the bladder to remove any NMIBC or MIBC.
* Has received a live or live attenuated vaccine within 30 days before the first dose of study intervention.
* Has a diagnosis of immunodeficiency or has a known history of human immunodeficiency virus (HIV) infection, Hepatitis B infection or known active Hepatitis C infection.
* Has a known psychiatric or substance abuse disorder.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | Up to approximately 60 months
  EFS is defined as the time from randomization to the first occurrence of any of the following events: progression of disease that precludes RC surgery; failure to undergo RC surgery in participants with residual disease and any radiographical disease present; gross residual disease left behind at the time of surgery; local or distant recurrence based on investigator assessments and/or biopsy, or death due to any cause.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to approximately 72 months
  pCR rate is defined as the percentage of participants having pCR. pCR is defined as absence of viable tumor (pT0N0) in examined tissue from RC and PLND, as assessed by blinded independent central review (BICR).
Overall Survival (OS) | Up to approximately 72 months
  Overall survival is defined as the time from randomization to death due to any cause.
Disease-Free Survival (DFS) | From approximately 20 weeks up to approximately 72 months
  DFS is defined as the time from post-surgery baseline scan until the first occurrence of either local or distant recurrence as assessed by investigator by CT or MRI and/or computerized tomography (CT) or magnetic resonance imaging (MRI) and or biopsy or death from any cause.
Pathologic Downstaging (pDS) Rate | Up to approximately 72 months
  pDS rate is defined as the percentage of participants having pDS. pDS is defined as participants with a tumor classification of <pT2 (includes pT0, pTis, pTa, pT1) and N0 in examined tissue from RC plus PLND as assessed by BICR.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 72 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 12 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Who Experienced Perioperative Complications | Up to approximately 12 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Change in Patient-Reported Outcomes from Baseline in Total Score of Functional Assessment of Cancer Therapy - General (FACT-G) | Baseline, Up to approximately 72 months
  The FACT-G is a health-related quality of life (HRQoL) 27-item questionnaire in patients being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 to 4, with higher scores indicating higher HRQoL. The total score can range from 0 to 108.
Change in Patient-Reported Outcomes from Baseline in Total Score of FACT-Bladder- (FACT-BI-Cys) | Baseline, Up to approximately 72 months
  Total Score of FACT BI-Cys is the sum of FACT-G total score and FACT-Bl-Cys score. FACT-Bl-Cys contains 17 items on the bowel, bladder, and sexual symptoms following cystectomy. The FACT-G is a health-related quality of life (HRQoL) 27-item questionnaire in patients being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 to 4, with higher scores indicating higher HRQoL. The total score of FACT-Bl-Cys can range from 0 to 168.
Change in Patient-Reported Outcomes from Baseline in FACT-BI-Cys-Trial Outcome Index (TOI) | Baseline, Up to approximately 72 months
  FACT-Bl-Cys Trial Outcome Index (TOI) is the sum of FACT-G PWB score, FWB score, and FACT-Bl-Cys score. FACT-Bl-Cys contains 17 items on the bowel, bladder, and sexual symptoms following cystectomy. The FACT-G is a health-related quality of life (HRQoL) 27-item questionnaire in patients being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0 to 4, with higher scores indicating higher HRQoL. The total score of FACT-Bl-Cys TOI can range from 0 to 116.
Change in Patient-Reported Outcomes from Baseline in EuroQol Five-Dimensional Questionnaire (EQ-5D-5L) Visual Analog Score (VAS) | Baseline, Up to approximately 72 months
  The EQ-5D-5L is a standardized instrument for use as a measure of health outcome. In the EQ-5D-5L VAS, the participant rates his or her general state of health at the time of the assessment on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time to Deterioration (TTD) in the Total Score of FACT-G | Up to approximately 72 months
  The FACT-G is a health-related quality of life (HRQoL) 27-item questionnaire in patients being treated for cancer. The FACT-G subscales include Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB). All items are scored on a 5-point Likert scale of 0-4, with higher scores indicating higher HRQoL. TTD is defined as the time from baseline to the first onset of patient-reported outcomes (PRO) deterioration. For the FACT-G questionnaire, deteriorations are defined as a decrease of 7 points or more (out of 108) from baseline in total score.
TTD in EQ-5D-5L VAS | Up to approximately 72 months
  The EQ-5D-5L is a standardized instrument for use as a measure of health outcome and includes 5 health state dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In the EQ-5D-5L VAS, the participant rates his or her general state of health at the time of the assessment on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. TTD is defined as the time from baseline to the first onset of PRO deterioration. For the EQ 5D-5L, deterioration is defined as a decrease of 7 points or more from baseline in the VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (175):
- United States (24):
  - Scripps MD Anderson ( Site 0010), La Jolla, California
  - Providence Saint John's Health Center ( Site 0075), Santa Monica, California
  - Georgetown University Medical Center ( Site 0022), Washington D.C., District of Columbia
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlando ( Site 0005), Orlando, Florida
  - Parkview Cancer Institute ( Site 0077), Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 0004), Indianapolis, Indiana
  - Ochsner Medical Center ( Site 0049), New Orleans, Louisiana
  - New England Cancer Specialists ( Site 0070), Scarborough, Maine
  - UMass Memorial Medical Center ( Site 0051), Worcester, Massachusetts
  - Henry Ford Hospital ( Site 0039), Detroit, Michigan
  - Mercy Hospital Saint Louis ( Site 0064), St Louis, Missouri
  - Morristown Medical Center ( Site 0015), Morristown, New Jersey
  - UNM Comprehensive Cancer Center-Clinical Research Office ( Site 0045), Albuquerque, New Mexico
  - New York University Perlmutter Cancer Center ( Site 0008), New York, New York
  - University Hospitals Cleveland Medical Center ( Site 0038), Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0021), Tulsa, Oklahoma
  - Portland VA Medical Center ( Site 0084), Portland, Oregon
  - Allegheny General Hospital ( Site 0048), Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center ( Site 0063), Houston, Texas
  - Central Texas Veterans Healthcare System ( Site 0057), Temple, Texas
  - Inova Schar Cancer Institute ( Site 0007), Fairfax, Virginia
  - Northwest Medical Specialties, PLLC ( Site 0061), Puyallup, Washington
  - Seattle Cancer Care Alliance/Univ of Washington Medical Center ( Site 0033), Seattle, Washington
  - Charleston Area Medical Center ( Site 0023), Charles Town, West Virginia
- Australia (5):
  - Mid North Coast Cancer Institute ( Site 1256), Port Macquarie, New South Wales
  - Southside Cancer Care Centre ( Site 1252), Sydney, New South Wales
  - Cairns Base Hospital ( Site 1257), Cairns, Queensland
  - Eastern Health ( Site 1255), Box Hill, Victoria
  - Peninsula Health Frankston Hospital ( Site 1258), Frankston, Victoria
- Belgium (5):
  - UZ Brussel ( Site 0358), Brussels, Bruxelles-Capitale, Region de
  - Jessa Ziekenhuis ( Site 0360), Hasselt, Limburg
  - CHU UCL Namur Site de Godinne ( Site 0354), Yvoir, Namur
  - O.L.V. Ziekenhuis Aalst ( Site 0356), Aalst, Oost-Vlaanderen
  - AZ Maria Middelares Gent ( Site 0353), Ghent, Oost-Vlaanderen
- Canada (8):
  - Tom Baker Cancer Centre ( Site 0100), Calgary, Alberta
  - Nova Scotia Health Authority ( Site 0109), Halifax, Nova Scotia
  - Kingston Health Sciences Centre ( Site 0103), Kingston, Ontario
  - Lakeridge Health ( Site 0104), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 0110), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0107), Toronto, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0105), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- Denmark (3):
  - Rigshospitalet University Hospital ( Site 0401), Copenhagen, Capital Region
  - Herlev og Gentofte Hospital. ( Site 0402), Herlev, Capital Region
  - Odense Universitetshospital ( Site 0403), Odense, Region Syddanmark
- France (12):
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0456), Bordeaux, Aquitaine
  - Centre Leon Berard ( Site 0465), Lyon, Auvergne
  - Centre Francois Baclesse ( Site 0459), Caen, Calvados
  - Centre Armoricain de Radiotherapie Imagerie medicale et Oncologie ( Site 0457), Plérin, Cotes-d Armor
  - Hopital Foch ( Site 0483), Suresnes, Hauts-de-Seine
  - CHU de Montpellier - Hopital Saint-Eloi ( Site 0469), Montpellier, Languedoc-Roussillon
  - Institut de Cancerologie de l Ouest Site Paul Papin ( Site 0453), Angers, Maine-et-Loire
  - Hopital Robert Schuman ( Site 0452), Metz, Moselle
  - Centre Jean Perrin ( Site 0460), Clermont-Ferrand, Puy-de-Dome
  - Clinique Victor Hugo ( Site 0463), Le Mans, Sarthe
  - CHU de Rouen ( Site 0493), Rouen, Seine-Maritime
  - Institut Sainte Catherine ( Site 0454), Avignon, Vaucluse
- Germany (7):
  - Klinikum der Eberhard-Karls-Universitaet Tuebingen ( Site 0502), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 0505), Erlangen, Bavaria
  - Universitaetsklinikum Carl Gustav Carus ( Site 0519), Dresden, Saxony
  - Universitaetsklinikum Magdeburg A.o.R. ( Site 0516), Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein-Campus Lubeck ( Site 0512), Lübeck, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin ( Site 0515), Berlin
  - Vivantes Klinikum am Urban ( Site 0522), Berlin
- Hungary (7):
  - Pecsi Tudomanyegyetem AOK ( Site 1009), Pécs, Baranya
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 1010), Szeged, Csongrád megye
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 1002), Szolnok, Jász-Nagykun-Szolnok
  - Bajcsy Zsilinszki Korhaz es Rendelointezet ( Site 1001), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 1006), Debrecen
  - Petz Aladar Megyei Oktato Korhaz ( Site 1012), Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 1007), Kaposvár
- Ireland (3):
  - Cork University Hospital ( Site 0722), Cork
  - Tallaght University Hospital ( Site 0710), Dublin
  - University Hospital Waterford ( Site 0723), Waterford
- Israel (10):
  - Ha Emek Medical Center ( Site 0808), Afula
  - Soroka Medical Center ( Site 0806), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0802), Haifa
  - Shaare Zedek Medical Center ( Site 0809), Jerusalem
  - Hadassah Ein Kerem Medical Center ( Site 0810), Jerusalem
  - Meir Medical Center ( Site 0803), Kfar Saba
  - Rabin Medical Center ( Site 0804), Petah Tikva
  - Sheba Medical Center ( Site 0801), Ramat Gan
  - Sourasky Medical Center ( Site 0807), Tel Aviv
  - Yitzhak Shamir Medical Center ( Site 0805), Ẕerifin
- Italy (8):
  - Policlinico Gemelli di Roma ( Site 0558), Roma, Abruzzo
  - Policlinico di Modena ( Site 0553), Modena, Emilia-Romagna
  - A.O.U. Policlinico Vittorio Emanuele - Presidio Gaspare Rodolico ( Site 0559), Catania
  - Istituto Nazionale Studio e Cura dei Tumori ( Site 0551), Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori ( Site 0552), Napoli
  - Fondazione Salvatore Maugeri IRCCS. ( Site 0554), Pavia
  - Azienda Ospedaliera San Camillo Forlanini ( Site 0560), Roma
  - Azienda Ospedaliera Santa Maria Terni ( Site 0557), Terni
- Japan (15):
  - Hirosaki University Hospital ( Site 1502), Hirosaki, Aomori
  - National Cancer Center Hospital East ( Site 1504), Kashiwa, Chiba
  - Ehime University Hospital ( Site 1508), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 1501), Sapporo, Hokkaido
  - University of Tsukuba Hospital ( Site 1503), Tsukuba, Ibaraki
  - Yokosuka Kyosai Hospital ( Site 1509), Yokosuka, Kanagawa
  - Nara Medical University Hospital ( Site 1510), Kashihara, Nara
  - Saitama Medical University International Medical Center ( Site 1505), Hidaka, Saitama
  - Chiba Cancer Center ( Site 1506), Chiba
  - Harasanshin Hospital ( Site 1515), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 1513), Hiroshima
  - Nagano Municipal Hospital ( Site 1516), Nagano
  - Osaka Metropolitan University Hospital ( Site 1512), Osaka
  - Tokushima University Hospital ( Site 1514), Tokushima
  - Tokyo Medical and Dental University Hospital ( Site 1517), Tokyo
- Mexico (4):
  - Centro de Urologia Avanzada del Noreste S.A. de C.V. ( Site 0254), Monterrey, Nuevo León
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V. ( Site 0300), Aguascalientes
  - Centro Estatal de Cancerologia de Chihuahua ( Site 0253), Chihuahua City
  - Instituto Nacional de Cancerologia ( Site 0256), Tlalpan
- Poland (5):
  - Centrum Onkologii im.prof. F. Lukaszczyka w Bydgoszczy ( Site 1068), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego ( Site 1062), Wroclaw, Lower Silesian Voivodeship
  - Europejskie Centrum Zdrowia Otwock ( Site 1057), Otwock, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 1051), Warsaw, Masovian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 1060), Bielsko-Biala, Silesian Voivodeship
- Russia (12):
  - Clinic of Bashkortostan State Medical University ( Site 0869), Ufa, Baskortostan, Respublika
  - Ivanovo Regional Oncology Dispensary ( Site 0852), Ivanovo, Ivanovo Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0861), Krasnoyarsk, Krasnoyarsk Krai
  - Kursk Regional Clinical Oncology Dispensary ( Site 0854), Kursk, Kursk Oblast
  - FSBI ""United Hospital with Polyclinic"" of the Administrative Department of the President of the Ru, Moscow, Moscow
  - Central Clinical Hospital with outpatient Clinic ( Site 0856), Moscow, Moscow
  - Bayandin Murmansk Regional Clinical Hospital ( Site 0859), Murmansk, Murmansk Oblast
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 0857), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 0865), Omsk, Omsk Oblast
  - Leningrad Regional Oncology Center ( Site 0868), Saint Petersburg, Sankt-Peterburg
  - Clinical Hospital Saint Luka ( Site 0867), Saint Petersburg, Sankt-Peterburg
  - Saratov State Medical University n.a. V.I.Razumovskiy ( Site 0866), Saratov, Saratov Oblast
- South Korea (6):
  - National Cancer Center ( Site 1354), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 1356), Seongnam-si, Kyonggi-do
  - Korea University Anam Hospital ( Site 1351), Seoul
  - Seoul National University Hospital ( Site 1352), Seoul
  - Asan Medical Center ( Site 1355), Seoul
  - Samsung Medical Center ( Site 1353), Seoul
- Spain (9):
  - Hospital San Pedro de Alcantara ( Site 0654), Cáceres, Extremadura
  - H. de Gerona Dr. Josep Trueta ( Site 0651), Girona, Gerona
  - Hospital Universitario Ramon y Cajal ( Site 0660), Madrid, Madrid, Comunidad de
  - Hospital Universitario Quiron Madrid ( Site 0657), Pozuelo de Alarcón, Madrid, Comunidad de
  - Instituto Valenciano de Oncologia - IVO ( Site 0662), Valencia, Valenciana, Comunitat
  - Hospital del Mar ( Site 0653), Barcelona
  - Hospital Universitario San Carlos ( Site 0663), Madrid
  - Hospital Universitario La Paz ( Site 0661), Madrid
  - Hospital Nuestra Sra. de Valme ( Site 0658), Seville
- Sweden (3):
  - Laenssjukhuset Ryhov ( Site 1205), Jönköping, Jönköping County
  - Akademiska Sjukhuset ( Site 1201), Uppsala, Uppsala County
  - Cancercentrum ( Site 1204), Umeå, Västerbotten County
- Thailand (4):
  - Ramathibodi Hospital. ( Site 1451), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1452), Bangkok, Bangkok
  - Maharaj Nakorn Chiangmai Hospital ( Site 1453), Chiang Mai
  - Srinagarind Hospital ( Site 1454), Khon Kaen
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tıp Fakultesi ( Site 0911), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0910), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 0906), Istanbul
  - Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 0901), Istanbul
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi ( Site 0909), Konya
  - Sakarya Universitesi Tip Fakultesi ( Site 0913), Sakarya
  - Karadeniz Teknik Universitesi Tip Fakultesi Farabi Hastanesi ( Site 0904), Trabzon
- Ukraine (10):
  - Cherkasy Regional Oncology Dispensary ( Site 0959), Cherkasy, Cherkasy Oblast
  - Regional Oncological Hospital ( Site 0956), Dnipro, Dnipropetrovsk Oblast
  - Dnipropetrovsk City Multidiscipline Clinical Hosp. 4 of DRC ( Site 0951), Dnipro, Dnipropetrovsk Oblast
  - MI Dnipr Regional Clinical Hospital named after I.I. Mechnikov ( Site 0963), Dnipropetrovsk, Dnipropetrovsk Oblast
  - Reg. Clinical Center of Urology and Nephrology n.a. V. I. Shapoval ( Site 0969), Kharkiv, Kharkivs’ka Oblast’
  - CNPE "Regional Center of Oncology" ( Site 0958), Kharkiv, Kharkivs’ka Oblast’
  - National Cancer Institute of the MoH of Ukraine ( Site 0962), Kyiv, Kyivska Oblast
  - Lviv Regional Clinical Hospital ( Site 0955), Lviv, Lviv Oblast
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 0967), Lviv, Lviv Oblast
  - Kyiv City Clinical Oncology Center ( Site 0960), Kyiv
- United Kingdom (8):
  - Aberdeen Royal Infirmary ( Site 0708), Aberdeen, Aberdeen City
  - Torbay Hospital ( Site 0704), Torquay, Devon
  - Kent and Canterbury Hospital ( Site 0709), Canterbury, England
  - Lister Hospital ( Site 0715), Stevenage, Hertfordshire
  - The Royal Marsden Foundation Trust ( Site 0702), London, London, City of
  - Imperial College Healthcare NHS Trust ( Site 0721), London, London, City of
  - Norfolk & Norwich University Hospital NHS Foundation Trust ( Site 0725), Norwich, Norfolk
  - Royal Cornwall Hospital ( Site 0703), Truro

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Galsky MD, Hoimes CJ, Necchi A, Shore N, Witjes JA, Steinberg G, Bedke J, Nishiyama H, Fang X, Kataria R, Sbar E, Jia X, Siefker-Radtke A. Perioperative pembrolizumab therapy in muscle-invasive bladder cancer: Phase III KEYNOTE-866 and KEYNOTE-905/EV-303. Future Oncol. 2021 Aug;17(24):3137-3150. doi: 10.2217/fon-2021-0273. Epub 2021 May 19. PMID 34008425
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26320&tenant=MT_MSD_9011